CLINICAL TRIAL: NCT03327740
Title: A Prospective Observational Cohort Study to Monitor and Compare the Occurrence of Hypersensitivity Reaction and Hepatotoxicity in Patients Receiving Dolutegravir (With and Without Abacavir) or Other Integrase Inhibitors (With or Without Abacavir)
Brief Title: PRJ2203: Dolutegravir Post Authorization Safety Study (PASS)
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201177; PRJ2203 (Other: GSK)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: Hypersensitivity reactions (HSR); HIV; Dolutegravir
MeSH Terms: conditions — Infections; Hypersensitivity | interventions — abacavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Subjects on DTG based ARV with ABC: These are subjects who begin a DTG based ARV regimen that includes ABC
  Interventions: Drug: DTG based ARV regimen with ABC
- Subjects that start DTG based ARV regimen but without ABC: These are subjects who begin a DTG-based ARV regimen that does not contain ABC
  Interventions: Drug: DTG based ARV regimen without ABC
- Subjects on other integrase inhibitor based regimen with ABC: These are subjects who begin other integrase inhibitor based regimens (RAL and EGV) that contains ABC
  Interventions: Drug: RAL or EGV based ARV regimens with ABC
- Subjects on other integrase inhibitor based regimen but no ABC: These are subjects that start non-ABC containing RAL or EGV based regimens
  Interventions: Drug: RAL or EGV based regimens without ABC
- Subjects that start any other DTG based ARV regimen: These are subjects who begin any other DTG based ARV regimen that will include DTG as monotherapy or two-drug regimens
  Interventions: Drug: Any other DTG based ARV regimen as monotherapy

INTERVENTIONS:
Drug: DTG based ARV regimen with ABC — ARV regimens containing DTG and ABC
  Groups: Subjects on DTG based ARV with ABC
Drug: DTG based ARV regimen without ABC — DTG based ARV regimens that do not contain ABC
  Groups: Subjects that start DTG based ARV regimen but without ABC
Drug: RAL or EGV based ARV regimens with ABC — RAL or EGV based regimens containing ABC
  Groups: Subjects on other integrase inhibitor based regimen with ABC
Drug: RAL or EGV based regimens without ABC — RAL or EGV based ARV regimens that do not contain ABC
  Groups: Subjects on other integrase inhibitor based regimen but no ABC
Drug: Any other DTG based ARV regimen as monotherapy — Any other DTG based ARV regimens including DTG as monotherapy or two-drug regimens.
  Groups: Subjects that start any other DTG based ARV regimen

SUMMARY:
Dolutegravir (DTG) is recommended for both treatment-naïve and treatment-experienced, HIV infected adults and paediatric subjects aged 12 years and older and weighing at least 40 kg. One case of suspected DTG hypersensitivity (HSR) reaction from among over 1500 subjects exposed to the drug at the time of submission in 4Q2012, has been identified; this subject experienced a diffuse maculopapular rash with fever and elevated liver enzymes. Isolated rash was uncommon in the DTG programme with less than 1% of clinical trial subjects experiencing treatment related rash. The pharmacovigilance strategy for DTG and DTG-containing products is to implement a post-marketing risk management program to further quantify the risk of HSR and compare it to that of other integrase inhibitors, and to possibly determine associated risk factors. In addition, the post-authorization safety study will monitor and compare hepatotoxicity and severe skin rash following initiation of DTG or other integrase inhibitor (raltegravir (RAL) or elvitegravir (EGV) based antiretroviral regimens (ARV). Further to be able to distinguish the above symptoms and reactions caused by DTG or the other integrase inhibitor regimen from that of abacavir (ABC), known to cause hypersensitivity reaction, the integrase inhibitor groups will be compared in combinations with and without ABC. This five year-long safety study will be conducted through collaboration with EuroSIDA, a well established prospective observational cohort study of more than 18,200 subjects followed in 107 hospitals in 31 European countries, plus Israel and Argentina. This is a five year-long non-interventional prospective cohort study nested within the EuroSIDA study. The study population will include HIV positive subjects over the age of 16 years from EuroSIDA clinical sites, who are new users of DTG or other integrase inhibitors with and without ABC. Following initiation of DTG with ABC based antiretroviral regimen or DTG without ABC or regimens containing other integrase inhibitors (RAL, EGV) with or without ABC or any other DTG based ARV regimen as monotherapy or two-drug regimens, the study will aim to a) Monitor and compare hypersensitivity reaction, b) Monitor and compare hepatotoxicity, and c) Monitor and compare severe skin rash among all subjects discontinuing DTG or other integrase inhibitor regimens for any reason.

ELIGIBILITY:
Inclusion Criteria:

* New users of DTG or users of other integrase inhibitor regimens (RAL and EGV)

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV positive subjects over the age of 16 years from EuroSIDA clinical sites, who are new users of DTG or users of other integrase inhibitor regimens (RAL and EGV).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2014-09-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with occurrence of hypersensitivity reactions (HSR), of any grade | Up to 5 years
  Hypersensitivity reactions including fever, rash, gastrointestinal symptoms, constitutional symptoms, respiratory symptoms and eosinophilia will be summarized.
Number of subjects with hepatic dysfunction | Up to 5 years
  Hepatic dysfunction will be indicated by liver chemistry tests

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare